CLINICAL TRIAL: NCT02526212
Title: Buprenorphine Group Medical Visits for Drug Users at Risk for HIV
Brief Title: Buprenorphine Group Medical Visits in Primary Care
Acronym: G-BMT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Aaron D. Fox, Assistant Professor of Medicine, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-3580; R34DA039041 (NIH)
Record Dates: First submitted 2015-07-24; First posted 2015-08-18 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Opioid-Related Disorders
Keywords: opioid use disorder; group counseling; office-based buprenorphine treatment
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Therapeutics; Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- G-BMT, Buprenorphine (Experimental): This arm will receive the G-BMT intervention, which will include group visits where 5-10 patients simultaneously receive care from a multidisciplinary team of a generalist physician and a behavioral specialist. The G-BMT intervention will last 90 minutes and include: BMT education, instruction on self-management skills, peer support, and individual medical management.
  Interventions: Behavioral: G-BMT; Drug: Buprenorphine
- Treatment as usual, Buprenorphine (Active Comparator): Primary care physicians who prescribe buprenorphine will be trained to follow a protocol of BMT intensification, which includes increased visit frequency, referral for mental health counseling, and referral to addiction treatment specialist.
  Interventions: Behavioral: Treatment as usual; Drug: Buprenorphine

INTERVENTIONS:
Behavioral: G-BMT — The G-BMT intervention will include weekly group visits (for 8 weeks) where 5-10 patients simultaneously receive care from a multidisciplinary team of a generalist physician and a behavioral specialist. Group visits will last 90 minutes and include: BMT education, instruction on self-management skills, peer support, and individual medical management.
  Other Names: Group Buprenorphine Maintenance Treatment (G-BMT)
  Arms: G-BMT, Buprenorphine
Behavioral: Treatment as usual — Primary care physicians who prescribe buprenorphine will be trained to follow a protocol of BMT intensification, which includes increased visit frequency, referral for mental health counseling, and referral to addiction treatment specialist.
  Arms: Treatment as usual, Buprenorphine
Drug: Buprenorphine — All participants will continue to receive maintenance treatment with buprenorphine-naloxone
  Other Names: Buprenorphine Maintenance Treatment (BMT)

SUMMARY:
The primary goal of this research is to improve the effectiveness of buprenorphine maintenance treatment (BMT) within primary care.

Investigators propose that providing BMT as part of a group medical visit (instead of an individual visit) will improve treatment outcomes for patients with persistent opioid abuse, because members become accountable to the group, are exposed to beneficial habits of others (i.e. positive deviance), and can receive efficacious behavioral interventions concomitantly with medical management

DETAILED DESCRIPTION:
Investigators have developed a preliminary model of BMT group medical visits, conducted focus groups with BMT patients and providers, and will use this data to develop a manualized group-based BMT intervention (G-BMT). Investigators will then conduct a randomized controlled trial (RCT) of the G-BMT intervention within primary care to preliminarily test its efficacy, acceptability, and feasibility. Participants who have persistent opioid abuse while receiving BMT in primary care will be randomized to the G-BMT intervention (40 participants in 5 groups) or to intensify BMT (treatment as usual) with their individual primary care physician (40 participants).

Hypothesis: In a 16-week RCT of G-BMT, participants who receive the G-BMT intervention (vs. treatment as usual) will have higher abstinence rates (primary outcome, efficacy), fewer HIV risk behaviors (efficacy), and greater satisfaction with treatment (acceptability) and adherence to medical visits (feasibility).

ELIGIBILITY:
Inclusion Criteria:

1. Currently receiving BMT at Montefiore community health center (CHC).
2. Received BMT for 12 or more weeks.
3. Persistent opioid abuse (positive toxicology for an unprescribed opioid at most recent test or in 50% or more of collected tests in the previous 6 months.)
4. Fluent in English of Spanish

Exclusion Criteria:

1) Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron D Fox, MD, MS, Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine
Locations (1):
- Comprehensive Health Care Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | G-BMT, Buprenorphine | Treatment as Usual, Buprenorphine
Started | 10 | 8
Completed | 8 | 7
Not Completed | 2 | 1
Not completed — Incarceration | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | G-BMT, Buprenorphine | Treatment as Usual, Buprenorphine | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54.5 [39 to 60] | 50.5 [43 to 54] | 52 [39 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 9 | 8 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 9 | 8 | 17
  Non-Hispanic Black | 1 | 0 | 1
  Non-Hispanic White | 0 | 0 | 0
Education [Count of Participants; unit: Participants] — College = completed some college or graduated
  Participants
    High School | 6 | 6 | 12
    College | 4 | 2 | 6
Housing Status [Count of Participants; unit: Participants] — Unstable housing = homeless, shelter, single-room occupancy hotel, living with friend or family
  Participants
    Unstable Housing | 6 | 6 | 12
    Rental Apartment | 4 | 2 | 6
Recent Incarceration [Count of Participants; unit: Participants] — Spent one or more day in jail or prison in the 90 days before enrollment
  Participants | 2 | 1 | 3
Unemployed [Count of Participants; unit: Participants] | 8 | 7 | 15
Parole [Count of Participants; unit: Participants] | 2 | 1 | 3
Alcohol use [Count of Participants; unit: Participants] — Reported alcohol use on at least one day in 30 days before enrollment
  Participants | 4 | 2 | 6
Heroin use [Count of Participants; unit: Participants] — Reported heroin use on at least one day in 30 days before enrollment
  Participants | 8 | 6 | 14
Any illicit opioid use [Count of Participants; unit: Participants] — Reported use of heroin, non-prescribed methadone, or non-prescribed opioid analgesics on at least one day in 30 days before enrollment
  Participants | 8 | 7 | 15
Cocaine use [Count of Participants; unit: Participants] — Reported cocaine use on at least one day in 30 days before enrollment
  Participants | 4 | 2 | 6
Injection drug use [Count of Participants; unit: Participants] — Reported injection drug use on at least one day in 30 days before enrollment
  Participants | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Opioid Abstinence at 8 Weeks
Description: Opioid abstinence will be based on self-reported opioid use in the prior 30 days at the 8 week visit and the results of urine toxicology test at the 8 week visit. Abstinence (yes) will require no self-reported opioid use and negative urine toxicology test for opiates, methadone, and oxycodone.
Time Frame: 8 weeks
Population: Intention to treat analysis - missing urine drug toxicology tests are considered to be positive for illicit opioids
Measure: Count of Participants; unit: Participants
Arm/Group | G-BMT, Buprenorphine | Treatment as Usual, Buprenorphine
Number analyzed (Participants) | 10 | 8
Participants | 0 | 1
Statistical Analysis 1: Comparison: G-BMT, Buprenorphine vs Treatment as Usual, Buprenorphine; Due to the small sample size, planned analyses that assessed for clustering by group assignment or primary care physician could not be conducted. Chi square using fisher's exact test was conducted to investigate differences in abstinence between study arms; Test type: Superiority; p = 0.44, Fisher Exact

2. Secondary Outcome: Number of Participants Who Were Retained in Buprenorphine Treatment at 3 Months and 6 Months
Description: Retention is defined as having a medical visit or active buprenorphine prescription 12-16 weeks (3 month retention) and 24-28 weeks (6 month retention) after protocol initiation.
Time Frame: 3 months, 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | G-BMT, Buprenorphine | Treatment as Usual, Buprenorphine
Number analyzed (Participants) | 10 | 8
Participants
  3 month retention | 8 | 7
  6 month retention | 8 | 6

3. Secondary Outcome: Number of Participants Who Reported Sharing Injection Equipment at 8 Weeks
Description: We used the HIV risk measure from the NIDA Seek, Test, Treat, and Retain for Vulnerable Populations study. Items for sexual risk behavior are from the Women's Health CoOp Baseline Questionnaire. Items for injection risk behavior are from the STTR Criminal Justice instrument. We will report the number of participants reporting sharing of injection equipment at 8 weeks following enrollment.
Time Frame: 8 weeks
Population: 8 week data missing for 4 participants in G-BMT arm and 3 participants in the treatment as usual arm
Measure: Count of Participants; unit: Participants
Arm/Group | G-BMT, Buprenorphine | Treatment as Usual, Buprenorphine
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

4. Secondary Outcome: Acceptability (Scale)
Description: Satisfaction with BMT will be measured on a 5-point Likert scale for participants following completion of the intervention. We used 17 items from the Primary Care Buprenorphine Satisfaction Scale. Each item addressed satisfaction with a specific component of buprenorphine treatment, which participants rated on a scale from 1 (very unsatisfied) to 5 (very satisfied). A higher score indicates greater satisfaction.
Time Frame: 16 weeks
Population: Acceptability data missing for 4 participants in G-BMT arm and 3 participants in the treatment as usual arm
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | G-BMT, Buprenorphine | Treatment as Usual, Buprenorphine
Number analyzed (Participants) | 6 | 6
units on a scale | 4.6 (0.29) | 4.8 (0.19)
Statistical Analysis 1: Comparison: G-BMT, Buprenorphine vs Treatment as Usual, Buprenorphine; Each of the 17 items were rated on a scale from 1 to 5. For each participant, the scores from these items were summed and divided by 17 for an average satisfaction score. The average satisfaction score was compared between study arms; Test type: Superiority; p = 0.20, t-test, 2 sided

5. Secondary Outcome: Feasibility (Percentage of Visits Attended)
Description: Visit adherence will be measured as the number of buprenorphine visits attended divided by the number of buprenorphine visits required per protocol and multiplied by 100 to give a percentage
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of visits attended
Arm/Group | G-BMT, Buprenorphine | Treatment as Usual, Buprenorphine
Number analyzed (Participants) | 10 | 8
percentage of visits attended | 69 [13 to 88] | 71 [29 to 100]

ADVERSE EVENTS:
Time Frame: Medical record review was conducted after 24 weeks had elapsed following enrollment.
Arm/Group | G-BMT, Buprenorphine | Treatment as Usual, Buprenorphine
All-Cause Mortality (participants affected / at risk) | 0/10 | 1/8
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 0/10 | 0/8

LIMITATIONS AND CAVEATS:
Due to the small sample size, several analyses were not conducted as planned. Narrow inclusion criteria limited recruitment. Though efficacy data is limited, this pilot study did provide useful information about group feasibility and acceptability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-16): https://cdn.clinicaltrials.gov/large-docs/12/NCT02526212/Prot_SAP_000.pdf